CLINICAL TRIAL: NCT03889145
Title: A Randomized, Open-label, Single Dose, 3-way Crossover Study to Evaluate the Drug-drugs Interaction Between Telmisartan, Amlodipine and Hydrochlorothiazide in Healthy Male Volunteers
Brief Title: A Study to Evaluate the Drug-drug Interaction Between Telmisartan, Amlodipine and Hydrochlorothiazide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID-TAH-1301
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telmisartan, Amlodipine (Active Comparator)
  Interventions: Drug: Telmisartan 80mg; Drug: Amlodipine10mg
- Hydrochlorothiazide (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide
- Telmisartan, Amlodipine, Hydrochlorothiazide (Experimental)
  Interventions: Drug: Telmisartan 80mg; Drug: Amlodipine10mg; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan 80mg — Telmisartan 80mg
  Arms: Telmisartan, Amlodipine; Telmisartan, Amlodipine, Hydrochlorothiazide
Drug: Amlodipine10mg — Amlodipine 10mg
  Arms: Telmisartan, Amlodipine; Telmisartan, Amlodipine, Hydrochlorothiazide
Drug: Hydrochlorothiazide — Hydrochlorothiazide 25mg
  Arms: Hydrochlorothiazide; Telmisartan, Amlodipine, Hydrochlorothiazide

SUMMARY:
A randomized, open-label, single dose, 3-way crossover study to evaluate the drug-drugs interaction between Telmisartan, Amlodipine and Hydrochlorothiazide in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 20 to 55 years
* Subjects who have 17.5 ~ 30.5 kg/m2 body mass index (BMI) and body weight that is more than 55kg
* Subjects who have no congenital or chronic disease within the last 3 years and have no pathological symptoms or findings as a result of medical examination.
* Suitable subject who is determined by laboratory tests such as hematology tests, blood chemistry, urinalysis test according to the characteristics of the drug and screening tests such as electrocardiography(ECG) test.
* Subject who fully understand the clinical trials after in-depth explanation given prior to the clinical study, decided to join the clinical trials by their will and signed consent form which approved by Chonbuk National University Hospital Institutional Review Board(IRB).

Exclusion Criteria:

* Subjects who have a history of blood, kidneys, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurological or allergic diseases that is clinically significant (Except untreated asymptomatic seasonal allergies at the time of administration)
* Subjects who have a history of gastrointestinal disease or gastrointestinal surgery which can affect drug absorption.
* Subjects who drink Alcohol > 210g/week within 6 months prior to the screening.
* Subjects who involved in other clinical trials within two months before the first dose medication characters.
* Subjects who show Systolic Blood Pressure ≤100 or ≥150 mmHg or Diastolic Blood Pressure ≤60 or ≥100 mmHg at screening
* Subjects who had alcohol or drug abuse within one year before the screening
* Subjects who took medication of drug-metabolizing enzymes that are known to significantly induce or inhibit within 30 days
* Subjects who smoke 20 cigarettes or more a day
* Subjects who take medicine within 10 days before the first investigational product administration.
* Subject who done the whole blood donation within two months or component blood donation within 1 month within 1 month prior to the first dosing.
* Subject who can increase risk due to clinical test and administration of drugs or has severe grade / chronic medical, mental condition or abnormal laboratory result that may interfere with the analysis of test results.
* Subjects with serious history of hypersensitivity or allergy to investigational product.
* Subjects with severe hepatic impairment or Gallbladder Disease.
* Subject with hereditary angioedema or a history of angioedema when treated with ACE(Angiotensin-Converting enzyme) inhibitor or ARB(Angiotensin II Receptor Blocker) therapy
* Subjects who take combination medication with aliskiren in Diabetic patient or moderate to severe renal insufficient subjects (glomerular filtration rate<60mL/min/1.73m2)
* Subjects with severe hepatic impairment
* Subjects who have severe aortic stenosis
* Subjects with acute or severe renal failure
* Subjects with hyponatremia or hypokalemia
* Subjects with Addison's disease
* Subjects with hypercalcemia
* Subjects who have galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects who are unwilling or unable to comply with the Lifestyle guidelines described in this protocol
* Subject who are inadequate for this study to participate judged by investigator

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2014-02-19 (Actual); Study Completion 2014-02-19 (Actual)

PRIMARY OUTCOMES:
AUClast | Hour 0 (Pre-dose), Hour 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144(Total 19 points)]
Cmax | Hour 0 (Pre-dose), Hour 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144(Total 19 points)]

SECONDARY OUTCOMES:
AUCinf | Hour 0 (Pre-dose), Hour 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144(Total 19 points)]
Tmax | Hour 0 (Pre-dose), Hour 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144(Total 19 points)]

OTHER OUTCOMES:
t1/2 | Hour 0 (Pre-dose), Hour 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144(Total 19 points)]
CL/F | Hour 0 (Pre-dose), Hour 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144(Total 19 points)]

REFERENCES:
- [Derived] Moon SJ, Jeon JY, Yu KS, Kim MG. Pharmacokinetic Interaction Among Telmisartan, Amlodipine, and Hydrochlorothiazide After a Single Oral Administration in Healthy Male Subjects. Clin Ther. 2019 Nov;41(11):2273-2282. doi: 10.1016/j.clinthera.2019.08.020. Epub 2019 Sep 26. PMID 31564513